CLINICAL TRIAL: NCT04948619
Title: Immune Function and Response to Vaccination Following Completion of Cancer Directed Systemic Therapy in Pediatric Patients With Cancer
Brief Title: Immune Function and Response to Vaccination After Cancer Therapy in Pediatric Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00081757; 00053603 (Other: Advarra IRB); LCI-PED-NOS-VACC-001 (Other: Atrium Health)
Record Dates: First submitted 2021-06-15; First posted 2021-07-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer
Keywords: Pediatric Oncology; Vaccine
MeSH Terms: conditions — Neoplasms | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Single booster vaccines (Other): Those subjects randomized to Arm A, single dose vaccine boosters, will receive non live vaccine boosters at the 3 month visit. Boosters for live vaccines will be given at the 6 month visit. Boosters will only be given as applicable for low titers tested at the baseline assessment visit. Subjects who have negative/undetectable titers to any vaccine at the 24 month visit will receive boosters to each applicable vaccine.
  Interventions: Biological: Vaccine
- Arm B - Staged revaccination series (Other): Those subjects randomized to Arm B, the full revaccination series, will receive applicable vaccines when titers are low (below normal range) at baseline. When indicated, non-live vaccines will be given at the 3, 6, and 9 month visits, live vaccines will be given at the 6 and 9 month visit. Subjects who have negative/undetectable titers to any vaccine at the 24 month visit will receive boosters to each applicable vaccine.
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Patients will have lab evaluations for immune function at baseline, 3, 6, 9 and 24 months post completion of treatment. At 3 months off therapy, patients with abnormal vaccine antibody titers will be randomized to receive either single booster vaccines or to begin a full revaccination series that models post-hematopoietic stem cell transplant vaccination strategies.

SUMMARY:
Pediatric cancer survivors have increased infection-related morbidity and mortality. This study will evaluate immune dysfunction following cancer directed systemic therapy completion, with attention to clinical relevance and infection rate in this population compared to healthy siblings, when applicable. The investigators will also restart vaccinations at earlier time points than previously studied, at 3 months post therapy, and will assess whether boosters or revaccination schedules are superior for regaining immunity against potentially serious infections in survivors.

DETAILED DESCRIPTION:
This study is a prospective, randomized trial. The target population is all patients between the ages of 2 and 21 years of age who complete cancer directed systemic therapy for any malignant diagnosis at our center over a 2 to 3-year time frame. The study will be conducted in the various disease-specific off therapy and survivorship clinics of Levine Children's Cancer and Blood Disorders. Patients will have lab evaluations for immune function at baseline, 3, 6, 12, and 24 months from last dose of cancer directed systemic therapy. At 3 months from last dose of cancer directed systemic therapy, patients with abnormal vaccine antibody titers will be randomized to receive either single booster vaccines or to begin a full revaccination series that models post-hematopoietic stem cell transplant vaccination strategies. Vaccines given will be directed against Haemophilus influenza type B, tetanus, diphtheria, pertussis, polio, hepatitis B, Streptococcus pneumoniae, measles, mumps, rubella, and varicella. Live vaccines (measles, mumps, rubella, and varicella) will be given at 6 months from last dose of cancer directed systemic therapy. Repeat vaccine antibody titers will be assessed at follow up visits as above to determine if there are differences in immediate or maintained immunity based on vaccine strategy used. For subjects <18 years of age, we will present health questionnaires to their caregiver to answer at each of the time points. Subjects ≥18 years of age will complete their own health questionnaire. These questionnaires will assess frequency, type, and severity of viral and bacterial infections requiring antibiotics in study patients and their closest healthy sibling in age, when applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, HIPAA authorization for release of personal health information, and assent, when applicable from the subject, parent, or legal guardian.
2. Age greater than or equal to 2 years and less than 22 years at the time of consent
3. Lansky/Karnofsky Performance Status of greater than 50 (ECOG less than 2) within 30 days prior to date of enrollment
4. Histological or cytological confirmation of any malignancy treated by the Pediatric Oncology team of Levine Children's Hospital
5. History of any malignant diagnosis treated with at least one cycle of cancer directed systemic therapy
6. Must be no more than 60 days from last dose of cancer directed systemic therapy at time of enrollment
7. As determined by the enrolling physician, ability of the subject and parent/caregiver to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

1. Malignant disease treated with observation, surgery, or radiotherapy alone
2. Known coexisting immunodeficiency
3. Subjects with normal baseline titers for all investigated vaccines
4. Known pregnancy
5. Documented previous severe allergic reaction to any vaccine or component of a vaccine
6. Documented current/active, severe infection, as determined by the investigator

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Vaccination comparison via objective lab measurements of vaccine titers | 2 years
  To compare single booster vaccination (Arm A) to full revaccination (Arm B) in terms of immune response at 24 months post cancer directed systemic therapy in pediatric subjects who have received cancer directed systemic therapy for any malignancy.

SECONDARY OUTCOMES:
Vaccine comparison at 12 & 24 months | Up to 2 years
  To compare single booster vaccination to full revaccination in pediatric subjects who have received cancer directed systemic therapy for any malignancy in terms of the prevalence of immune abnormalities at 12 and 24 months completion.
Infection Rates | Up to 2 years
  Evaluate infection rates (over a 2-year post randomization period) between subjects with residual immune dysfunction versus subjects with recovered immune function
Healthy Sibling comparison | Up to 2 years
  Evaluate infection rates in enrolled subjects and compare to healthy siblings, when applicable
Immune Abnormalities - Malignancy | Up to 2 years
  Evaluate the prevalence of immune abnormalities at 12 and 24 months as a function of type of malignancy and length of treatment
Immune Abnormalities - Primary Vaccination Status | Up to 2 years
  Evaluate the prevalence of immune abnormalities as a function of primary vaccination status

OTHER OUTCOMES:
Safety - Potential Side Effects | Up to 5.5 years
  To summarize the rates of potential side effects thought by the investigator to be related to each vaccine strategy, including fever, rash, myalgias, injection site reaction, infection, or anaphylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Hinson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No